CLINICAL TRIAL: NCT03078972
Title: Effective Mechanical Circulatory Support on Exercise Capacity in Heart Failure
Brief Title: Effect of mechanIcal circulatoRy Support ON Exercise Capacity aMong pAtieNts With Heart Failure
Acronym: IRONMAN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1635
Record Dates: First submitted 2017-02-28; First posted 2017-03-14 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Approximately 20cc of blood will be collected during testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Advanced Heart Failure: 40 patients with advanced heart failure scheduled to undergo Left Ventricular Assist Device (LVAD) insertion will be recruited for testing. Test subjects will complete testing prior to, and following LVAD implantation.
- Healthy controls: 10 age-matched healthy individuals will be recruited to establish normal/reference values.
- Mild Heart Failure: A second control group comprised of 10 age-matched individuals will be recruited to establish normal/reference values for individuals with mild, medically managed heart failure.

SUMMARY:
This study will evaluate how the cardiovascular system interacts with mechanical hearts to provide blood flow to the body during exercise. Two aims are proposed: 1) to determine the impact of a mechanical heart on exercise pressor reflexes in heart failure patients; and 2) to define the primary determinant(s) of exercise capacity in heart failure patients before and after device implantation.

ELIGIBILITY:
Advanced Heart Failure-

Inclusion Criteria:

* Individuals with severely reduced left ventricular systolic function that are scheduled to undergo LVAD insertion

Exclusion Criteria:

* uncontrolled diabetes with peripheral neuropathy (interferes with acquisition of MSNA signal)
* Individuals with clinical right ventricular failure, defined as moderate-severely reduced RV systolic function on echocardiography, or clinical evidence of RV failure (elevated jugular venous pressures, significant peripheral edema)
* Individuals with moderate-severe preexisting aortic insufficiency, as these patients will typically undergo a Park stitch at time of CF-LVAD insertion to permanently close the aortic valve and prevent worsening aortic insufficiency; and
* Disorders that adversely influence exercise ability (e.g. arthritis, peripheral vascular disease, pulmonary disease)

Mild Heart Failure -

Inclusion Criteria:

* Individuals with medically managed left ventricular systolic function that are NOT scheduled to undergo LVAD insertion
* HF patients with ejection fraction <35-40%

Exclusion Criteria:

* Individuals requiring systemic anticoagulation with vitamin-K antagonists or new/direct oral anticoagulants ("NOAC"/"DOAC")
* Disorders that adversely influence exercise ability (e.g. arthritis, peripheral vascular disease, pulmonary disease)
* History of uncontrolled arrhythmias (e.g. ventricular tachycardia or nonsustained ventricular tachycardia).

Healthy Controls -

Inclusion Criteria:

- Persons without a past medical history of cardiovascular disease or related disease (e.g. hypertension, diabetes, peripheral vascular disease, arrhythmias, stroke/transient ischemic attack) and are not taking any cardiac-related medications (e.g. antihypertensive medications)

Exclusion Criteria:

* Individuals requiring systemic anticoagulation with vitamin-K antagonists or new/direct oral anticoagulants ("NOAC"/"DOAC")
* Disorders that adversely influence exercise ability (e.g. arthritis, peripheral ascular disease).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 - HF patients with advanced heart failure who are scheduled to undergo LVAD insertion (Advanced Heart Failure)
  10 - HF patients with mild heart failure who are not scheduled to undergo LVAD insertion, to serve as first control group (Mild Heart Failure)
  10 - Age-matched healthy individuals, with no past medical history, to serve as a second control group (Healthy Controls)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-04-07 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the sympathetic neural response. | 4 weeks prior to implantation and 6 months post implantation.
  The primary outcome will be the difference in the muscle sympathetic neural response (MSNA) to handgrip and post-exercise circulatory arrest (PECA) before and after Continuous-flow left ventricular assist device (CF-LVAD) insertion
Change in VO2. | 4 weeks prior to implantation and 6 months post implantation.
  The primary outcome will be the change in the VO2 (maximum rate of oxygen consumption) before and after CF-LVAD insertion.

SECONDARY OUTCOMES:
Changes in the hemodynamic response. | 4 weeks prior to implantation and 6 months post implantation.
  This outcome will evaluate any difference in the hemodynamic response (heart rate and blood pressure) to handgrip and PECA before and after CF-LVAD
VO2 relationship and ventilatory threshold (1) | 4 weeks prior to implantation and 6 months post implantation.
  Cardiac output (Qc): VO2 relationship and ventilatory threshold before and after CF-LVAD insertion.
VO2 relationship and ventilatory threshold (2). | 4 weeks prior to implantation and 6 months post implantation.
  Determinants of Qc after CF-LVAD insertion (ie, contribution from device v. contribution from left ventricle).
VO2 relationship and ventilatory threshold (3). | 4 weeks prior to implantation and 6 months post implantation.
  Qc, VO2, ventilatory threshold and exercise capacity at increased pump speed.
VO2 relationship and ventilatory threshold (4). | 4 weeks prior to implantation and 6 months post implantation.
  Bloodflow to the periphery, as measured by transcranial Doppler to assess brain bloodflow during exercise/activity.
Oxygen uptake and utilization | 4 weeks prior to implantation and 6 months post implantation.
  Cerebral and musculoskeletal oxygen uptake by near-infrared spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: William K Cornwell, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Snschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buchanan C, Buchanan C, Riordan M, Byrd J, Schulte M, Kohrt WM, Ambardekar AV, Allen LA, Wolfel G, Lawley J, Levine BD, Cornwell WK 3rd. Cardiopulmonary Performance Among Heart Failure Patients Before and After Left Ventricular Assist Device Implantation. JACC Heart Fail. 2024 Jan;12(1):117-129. doi: 10.1016/j.jchf.2023.06.017. Epub 2023 Aug 23. PMID 37632493
- [Derived] Edward JA, Parker H, Stohr EJ, McDonnell BJ, O'Gean K, Schulte M, Lawley JS, Cornwell WK 3rd. Exertional Cardiac and Pulmonary Vascular Hemodynamics in Patients With Heart Failure With Reduced Ejection Fraction. J Card Fail. 2023 Sep;29(9):1276-1284. doi: 10.1016/j.cardfail.2023.01.010. Epub 2023 Mar 5. PMID 36871613
- [Derived] Sailer C, Edelmann H, Buchanan C, Giro P, Babcock M, Swanson C, Spotts M, Schulte M, Pratt-Cordova A, Coe G, Beindorff M, Page RL 2nd, Ambardekar AV, Pal JD, Kohrt W, Wolfel E, Lawley JS, Tarumi T, Cornwell WK 3rd. Impairments in Blood Pressure Regulation and Cardiac Baroreceptor Sensitivity Among Patients With Heart Failure Supported With Continuous-Flow Left Ventricular Assist Devices. Circ Heart Fail. 2021 Jan;14(1):e007448. doi: 10.1161/CIRCHEARTFAILURE.120.007448. Epub 2021 Jan 19. PMID 33464953